CLINICAL TRIAL: NCT02713854
Title: Human Embryonic Stem Cell-derived Trophoblastic Spheroid (BAP-EB) as a Predictive Tool for Endometrial Receptivity and Pregnancy Outcome of in Vitro Fertilization Treatment
Brief Title: BAP-EB as a Predictive Tool for Endometrial Receptivity and Pregnancy Outcome of IVF Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The University of Hong Kong-Shenzhen Hospital (Other); Kwong Wah Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BAP-EB-2016-protocol-v1
Record Dates: First submitted 2016-03-09; First posted 2016-03-21 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2021-04

CONDITIONS: Subfertility
Keywords: Subfertility; In-vitro fertilization; BAP-EB; Endometrial epithelial cells; Repeated implantation failure
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endometrial biopsy group (Experimental): Women who have an endometrial biopsy 2-3 months prior to IVF
  Interventions: Procedure: endometrial biopsy

INTERVENTIONS:
Procedure: endometrial biopsy — An endometrial biopsy taken 2-3 months prior to IVF cycle

SUMMARY:
To determine the predictive value of attachment rate of human embryonic stem cells (hESC)-derived trophoblast spheroids (BAP-EB, embryo surrogate) onto endometrial epithelial cells (EEC) on success of IVF treatment and to use the model to identify EEC surface biomarkers for endometrial receptivity.

DETAILED DESCRIPTION:
Study Objectives and Purpose:

There are three objectives in this study:

1. To determine the predictive value of the attachment rate of BAP-EB onto EEC on success of IVF treatment. The attachment rate of BAP-EB onto EEC of subfertile women in a natural cycle preceding the IVF cycle will be determined and correlated with the cumulative live birth rate in a subsequent stimulated IVF cycle and the derived frozen-thawed embryo transfer (FET) cycles.
2. To identify the surface molecules on EEC responsible for attaching to BAP-EB. The biotin-labeled primary EEC surface proteins that bind onto BAP-EB will be purified and identified by mass spectrometry. The bound proteins from "receptive" and "non-receptive" endometrial cell lines will be compared. The expression of the surface proteins on endometrial samples obtained in Objective 1will be correlated with their BAP-EB attachment rate.
3. To compare the BAP-EB attachment rate and expression of the attachment-related "receptive" EEC surface molecules between pre-receptive and receptive endometrium and between women with repeated implantation failure (RIF) and subfertile women due to male factors. To identify women with endometrial defects, women with RIF and failed IVF after preimplantation genetic screening (PGS) will be recruited. The latter recruitment criterion excludes RIF due to embryo aneuploidy.

Subjects:

Patients will be recruited from the Centre of Assisted Reproduction and Embryology, the University of Hong Kong at Queen Mary Hospital (HKU-QMH CARE) and at University of Hong Kong-Shenzhen Hospital (HKU-SZH CARE), the Dr Stephen Chow Chun-kay Assisted Reproduction Centre, Kwong Wah Hospital (SCCARC).

Treatment of Subjects:

Endometrial biopsies will be collected from the subjects and the attachment rate of BAP-EB onto isolated EEC will be associated with the implantation and pregnancy outcomes in IVF and the expressions of the isolated surface proteins.

Study duration: 36 months

Assessment of Safety:

1. Specification of safety parameters. Abdominal pain after endometrial aspirate
2. The methods and timing for assessing, recording, and analysing safety parameters. Subjects will be asked to contact investigators if they notice abdominal pain after endometrial aspirate
3. Procedures for eliciting reports of and for recording and reporting adverse event and intercurrent illnesses. Any abdominal pain will be documented in subjects' medical notes and they will be asked for any adverse effects and intercurrent illness when receiving IVF treatment.
4. The type and duration of the follow-up of subjects after adverse events. Subjects will be followed up in the Department of Obstetrics and Gynaecology as long as they have the adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Subfertile women indicated for the first IVF or women with cryopreserved embryos at HKU-QMH CARE, HKU-SZH CARE and SCCARC
* Women indicated for IVF treatment with a normal uterine cavity as demonstrated by saline infusion sonogram or hysteroscopy
* Women with regular ovulatory cycles

Exclusion Criteria:

* The presence of an endometrial polyp or fibroid distorting the uterine cavity
* The presence of untreated hydrosalpinx
* IVF treatment carried out for preimplantation genetic diagnosis
* The use of donor oocytes

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-07-04 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Cumulative live birth rate | 36 months
  Cumulative birth rate: delivery of a live birth beyond 24 weeks of gestation in that episode of IVF treatment

SECONDARY OUTCOMES:
Clinical pregnancy | 6 weeks
  presence of at least one gestational sac on ultrasound at 6 weeks
Ongoing pregnancy | 20 weeks
  presence of at least one fetal heart pulsation on ultrasound beyond 20 weeks
Implantation rate | 6 weeks
  Number of ultrasound detected embryonic sacs divided by the number of embryos transferred.
Miscarriage rate | 20 weeks
  Number of miscarriages before 20 weeks divided by the number of women with a positive pregnancy test.
Multiple pregnancy | 6 weeks
  A pregnancy with more than one gestational sac detected on ultrasound at 6 weeks
Live birth rate | 42 weeks
  Live birth rate: delivery of a live birth beyond 24 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Ernest HY Ng, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Obstetrics and Gynaecology, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee YL, Ruan H, Lee KC, Fong SW, Yue C, Chen ACH, Lee KF, Lam MT, Yeung WSB, Li RHW, Ng EHY. Attachment of a trophoblastic spheroid onto endometrial epithelial cells predicts cumulative live birth in women aged 35 and older. Fertil Steril. 2023 Aug;120(2):268-276. doi: 10.1016/j.fertnstert.2023.03.013. Epub 2023 Mar 20. PMID 36940739